CLINICAL TRIAL: NCT00005389
Title: Effect of Drug Therapy on Reinfarction Risk in Women
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4295; R01HL053375 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2001-04

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Heart Diseases

SUMMARY:
To evaluate the safety of calcium-channel blockers in the secondary prevention of myocardial infarction in women.

DETAILED DESCRIPTION:
BACKGROUND:

Research on heart disease in the 196Os and 197Os was primarily concerned with risk factors for 'premature' atherosclerosis, which was most dramatically apparent in working middle-aged men who suffered heart attacks or died suddenly. This focus on 'premature' disease was an important initial step, but it resulted in a relative neglect of studies in older adults and in all women. Coronary heart disease remains nonetheless a major cause of morbidity and mortality among women.

Given the consistent findings from clinical trials that calcium-channel blockers administered following myocardial infarction do not decrease the risk of death or reinfarction, and that some drugs of this class may actually increase the risk, it is unlikely that future trials of this therapy in women will be conducted. Yet the calcium-channel blockers are used with increasing frequency in women following myocardial infarction. The only ethical method of conducting studies of the safety of these drugs in women is through observational studies. Data from the study can help to guide clinical practice and can assist in the design of appropriate secondary prevention trials in women.

DESIGN NARRATIVE:

On-going studies of hormone-replacement therapy in women at Group Health Cooperative of Puget Sound (GHC) identified all female enrollees who suffered a first heart attack since 1986; the study expanded this inception cohort through 1996. Information from medical record review and GHC databases were used to assess risk factors and co-morbid conditions, both at entry into the cohort and up to ten years of follow-up, and to identify recurrent cardiovascular events and deaths. A complete record of prescription drug exposure during the follow-up period was obtained for each subject from the GHC computerized pharmacy database. Although the main hypothesis related to reinfarction risk in women, men were studied as well to facilitate comparison of the results of this observational study with those of the clinical trials. According to conservative estimates of the available sample size, the investigators had 86 percent power to detect a relative risk of 1.45 in women alone, and 85 percent power to detect a relative risk of 1.25 in men and women combined, for the association of calcium-channel blocker use with fatal or non-fatal reinfarction. The study also examined the safety and efficacy of other cardiovascular drugs commonly used in women after myocardial infarction, including angiotensin converting-enzyme inhibitors, lipid-lowering drugs, and estrogen replacement therapy.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 1998-08

REFERENCES:
- [Background] Heckbert SR, Weiss NS, Koepsell TD, Lemaitre RN, Smith NL, Siscovick DS, Lin D, Psaty BM. Duration of estrogen replacement therapy in relation to the risk of incident myocardial infarction in postmenopausal women. Arch Intern Med. 1997 Jun 23;157(12):1330-6. PMID 9201007
- [Background] Kaplan RC, Heckbert SR, Weiss NS, Wahl PW, Smith NL, Newton KM, Psaty BM. Postmenopausal estrogens and risk of myocardial infarction in diabetic women. Diabetes Care. 1998 Jul;21(7):1117-21. doi: 10.2337/diacare.21.7.1117. PMID 9653605